CLINICAL TRIAL: NCT03914079
Title: Evaluation of the CAD-det System, a Novel Non-Invasive Acoustic Diagnostic for the Diagnosis of Coronary Artery Disease
Acronym: CAD-det
Status: Suspended | Type: Observational
Why Stopped: Sponsor due to COVID-19
Sponsor: AusculSciences Canada Inc. (Industry)
Collaborators: Ottawa Heart Institute Research Corporation (Other); Horizon Health Network (Other); University of Calgary (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: CAD-det-Research-Study
Record Dates: First submitted 2019-01-31; First posted 2019-04-16 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Cardiovascular Disease
Keywords: Coronary Artery Disease; Cardiovascular Disease; Atherosclerosis; Coronary Occlusion; Non-Invasive Medical Device; Cardiac Diagnostics
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Atherosclerosis; Coronary Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of this multi-center study is to collect and study the acoustic and electrical signals created by the heart during the cardiac cycle as a result of stenosis or plaque associated with coronary artery disease (CAD).

DETAILED DESCRIPTION:
This research intends to evaluate acoustic and electrical cardiovascular signals in patients with known or suspected CAD and establish the ability of the CAD-det System to accurately and reliably detect them utilizing coronary computed tomography (CCTA) and invasive coronary angiography (ICA) as reference standards. In addition, this study will collect clinical and acoustic data of other cardiac pathologies to better understand their impact on the acoustic signatures associated with CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years;
2. Suspected or known CAD;
3. Able and willing to comply with the study procedures;
4. Referred to ICA or CCTA for CAD characterization;
5. Willingness and ability to sign the Informed Consent Form.

Exclusion Criteria:

1. Unwillingness or inability to provide informed consent;
2. Age less than 19 years;
3. Pregnancy;
4. Skin injury/diseases/lesions that would preclude safe application of the CAD-det device.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 2,000 men and women age 19 and over with suspected or known CAD referred for clinically indicated Invasive Coronary Angiography (ICA) or Coronary Computed Tomography Angiography (CCTA).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants suspected of having Coronary Artery Disease | up to 1 Year
  Collection of all acoustic cardiac data to allow for the acoustic discrimination of the presence and degree of CAD in diseased and healthy participants.

SECONDARY OUTCOMES:
Estimation of coronary artery stenosis by the CAD-det device. | up to 1 year
  CAD-det results will be categorized by sex as:
  1. Acoustic and electrical signals consistent with 0-30% diameter stenosis (Negative for CAD);
  2. Acoustic and electrical signals consistent with 31-49% diameter stenosis (Pr-clinical / Negative);
  3. Acoustic and electrical signals consistent with 50-69% diameter stenosis (Positive);
  4. Acoustic and electrical signals consistent with 70% or greater diameter stenosis (Positive); and
  5. Equivocal or non-diagnostic.
Estimation of coronary artery stenosis by CCTA and ICA categorized by sex as: | up to 1 year
  1. 0 - 30% diameter stenosis (Negative);
  2. 31 - 49% diameter stenosis (Negative / Pre-clinical);
  3. 50 - 69% diameter stenosis (Positive);
  4. 70% or greater diameter stenosis (Positive); and
  5. Equivocal
  In cases where a participant undergoes both CCTA and ICA, the ICA results shall serve as the reference method results used for statistical analysis of the diagnostic accuracy of CAD-det. In participants with equivocal ICA and when invasive coronary physiology or functional assessments (eg. FFR, iFR, Pd/Pa, RFR) are performed, these assessments will be used to ascertain if the CAD-det can determine functional (hemodynamically significant) CAD.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chow, MD, FRCP(C), Principal Investigator — University of Ottawa Heart Institute (UOHI)
Locations (3):
- Canada (3):
  - Foothills Medical Centre (University of Calgary), Calgary, Alberta
  - Horizon Health Network, Saint John Regional Hospital, Saint John, New Brunswick
  - University of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makaryus AN, Makaryus JN, Figgatt A, Mulholland D, Kushner H, Semmlow JL, Mieres J, Taylor AJ. Utility of an advanced digital electronic stethoscope in the diagnosis of coronary artery disease compared with coronary computed tomographic angiography. Am J Cardiol. 2013 Mar 15;111(6):786-92. doi: 10.1016/j.amjcard.2012.11.039. Epub 2013 Jan 1. PMID 23290309
- See also: Study Sponsor — https://ausculsciences.com/